CLINICAL TRIAL: NCT05697068
Title: Tailored Behavioral Intervention to Prevent Household and Community Spread of COVID-19 Among Latinos
Brief Title: Intervention to Prevent Household and Community Spread of COVID-19 Among Latinos
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Family Health Centers of San Diego (Other)
Responsible Party: Principal Investigator, Noe Crespo, Associate Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MD016324 (NIH)
Record Dates: First submitted 2023-01-20; First posted 2023-01-25 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: SARS-CoV-2 Infection
Keywords: SARS-CoV-2; COVID-19; Prevention; Secondary Infection; Hispanics; Latinos; Household; Community; Clinic
MeSH Terms: conditions — COVID-19; Coinfection

STUDY DESIGN:
Intervention Model Description: Index patients will be randomly assigned (in real-time) to one of the two experimental groups using a predetermined randomization schedule (blocks of 40 randomly assigned numbers, stratified by study condition). Enrollment and randomization will be conducted in groups/waves of 40 index patients per wave. Enrollment and randomization will continue for each wave until 40 index patients have been randomized.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard-of-Care (Active Comparator): Patients who test positive will receive a call from the provider who conducted the test to notify them of the test result and provide standard-of-care counseling (e.g., health education, link them to resources). Index patients are entered into a COVID-19 patient registry in the Federally Qualified Health Center's electronic health record system (which also is linked to the clinic's COVID-19 dashboard) and monitored closely, with telemedicine follow-ups provided by skilled clinical staff every two-to-three days, and in-person follow-ups provided as needed.
  Interventions: Behavioral: COVID Prevention Program (CPP)
- Enhanced Standard-of-Care (Experimental): In addition to the aforementioned standard-of-care actions, index patients in the enhanced standard-of-care group will receive tailored phone/mobile counseling (motivational interviewing) focused on implementing strategies to prevent immediate household spread of COVID-19, followed by weekly text messaging for a total of 6 weeks.
  Interventions: Behavioral: COVID Prevention Program (CPP)

INTERVENTIONS:
Behavioral: COVID Prevention Program (CPP) — This project is a promotor/a-led COVID-19 Prevention Program (CPP) for Latino patients of a Federally Qualified Health Center (FQHC) who are recently diagnosed with SARS-CoV-2. The program will implement immediate risk reduction strategies to prevent household spread of COVID-19, followed by risk reduction strategies to prevent community spread. Patients and household members who agree to participate will be patients of the FQHC (the covered entity) and will have completed a broad consent that authorizes program activities (e.g., COVID-19 testing, individualized counseling). Patients are free to refuse to participate in the CPP without impact on other services they may receive at the clinic. Research activities will be managed by study's measurement team, which involves surveys conducted on index patients at baseline, 1-, 6-, 12-, and 24-months. Written informed consent will be obtained for all research activities occurring outside of clinical care.

SUMMARY:
This study will examine the effectiveness of a 6-week behavioral intervention for patients who are recently diagnosed with COVID-19. Patients and their households will be randomized to one of two groups (Standard of Care vs. Enhanced Standard of Care). Patients in the Standard-of-Care group will receive established clinical care and follow-up. Patients in the Enhanced Standard-of-Care group will receive standard-of-care plus tailored, real-time text messaging and virtual counseling delivered by promotores/as. The investigators hypothesize that households in the Enhanced Standard-of-Care group will have fewer (any new) household COVID-19 infectivity rates compared to households in the standard-of-care group post-intervention.

DETAILED DESCRIPTION:
The study team will develop and test a novel tailored behavioral intervention for patients of a Federally Qualified Health Center who are recently diagnosed with COVID-19. The study is a pragmatic, quality improvement randomized controlled trial (RCT). This research is looking to enroll 256 index patients and their households. Index patients and their households will be invited to participate in the COVID Prevention Program, which includes free COVID-19 testing for exposed household members. Index patients will be randomized to one of two groups: (a) the Standard-of-Care comparison group who will receive established clinical care and follow-up, or (b) the Enhanced Standard-of-Care group, who will receive standard-of-care plus tailored, real-time mobile/virtual counseling delivered by promotores/as. The intervention will use theory- and evidence-based strategies for behavior change and maximize the use of mobile phone applications and technologies to capture real-time behavioral, social, and contextual data (via Ecological Momentary Assessment). The intervention will utilize motivational interviewing techniques to tailor strategies to index patients' home environment/context and social/emotional needs. The intervention will target immediate risk of household spread, followed by risk of community spread. The primary outcome assessed will be a new positive antibody test within a household (post-baseline), as assessed by a blood draw collected by a certified phlebotomist. Secondary research outcomes will be assessed via self-report surveys. Surveys will include socioeconomic status indicators and demographics, as well as measures of mental health (e.g., depression), physical health (chronic conditions), health behaviors (social distancing, hand washing & wearing face covering), as well as comorbidities and risk factors for severe COVID-19 outcomes. Primary and secondary outcomes will be measured at 5 timepoints: baseline, 6-weeks, 6-months, 12-months, and 24-months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of a federally qualified health center (+18yrs)
* Test positive for COVID-19

Exclusion Criteria:

* Planning to move out of state in the next year
* Cognitive impairment that is contraindicated to receiving counseling and following behavioral strategies (e.g., schizophrenia, Down syndrome)
* Living in a transitionary home or homeless.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of households with SARS-CoV-2 Antibodies | Baseline & 1-, 6-, 12-, and 24-months post-baseline.
  Antibodies assessed by a blood draw collected by a certified phlebotomist. SARS-CoV-2 Nucleocapsid and Spike Protein IgG, used to accurately determine prior infection and/or vaccination.

SECONDARY OUTCOMES:
Number of households with SARS-CoV-2 Active Infection | Baseline, 3-5 days post-baseline, and 7-9 days post-baseline.
  Active infection assessed by self-administered anterior nasal swab. SARS-CoV-2 RT-PCR used to determine if exposed household member has been infected and/or can exit quarantine early.

OTHER OUTCOMES:
Number of participants with risk reduction behaviors | Baseline & 1-, 6-, 12-, and 24-months post-baseline.
  Secondary outcomes measured via self-report surveys. Surveys include socioeconomic status indicators and demographics, measures of mental health (e.g., depression), physical health (chronic conditions) and health behaviors (social distancing, hand washing & wearing face covering), comorbidities, and risk factors for severe COVID-19 outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Noe C Crespo, M.P.H, Ph.D., Principal Investigator — San Diego State University Research Foundation
Locations (1):
- San Diego State University Research Foundation, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crespo NC, Godino J, Behar A, Dionicio P, de la Torre CL, Fraga K, Santoscoy M, Elder JP, Oren E, Lin CD, Arredondo EM, Madanat H, Ramers CB. COVID Prevention Program: Rationale and methodology of a tailored behavioral intervention to prevent household and community spread of COVID-19 among Latinos. Contemp Clin Trials. 2025 Sep;156:108046. doi: 10.1016/j.cct.2025.108046. Epub 2025 Aug 13. PMID 40816435